CLINICAL TRIAL: NCT00677391
Title: Randomized Trial of Obese Non-Diabetic Malaysians Using Sibutramine: A Randomized Double-Blind Placebo-Controlled Study of Sibutramine in the Management of Obese Subjects in Malaysia
Brief Title: Efficacy and Safety Study of Sibutramine in Overweight Non-Diabetic Malaysian Population
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Peter Bacher, Global Project Head, Abbott
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MLAY-02-001
Record Dates: First submitted 2008-05-12; First posted 2008-05-14 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — sibutramine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Sibutramine
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sibutramine — Capsules, Wk 0: 10mg, once daily; Wks 4-24: 10mg or 15mg, once daily, dosage escalation based upon investigator's assessment.
  Other Names: ABT-991; Meridia; Reductil
  Arms: 1
Drug: Placebo — Capsules, once daily
  Arms: 2

SUMMARY:
The primary objective of this study was to evaluate the efficacy and the safety of sibutramine vs. placebo in combination with a hypocaloric diet on weight-loss in overweight and obese Malaysian subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject did not adequately respond (i.e., did not achieve or maintain > 5%weight loss) to an appropriate non-pharmacologic weight-reducing regimen (i.e., diet and exercise) within 3 months prior to Screening.
* The subject was male or female and between 18 and 65 years of age.
* The subject has nutritional obesity and BMI >= 27 kg/m2 associated with dyslipidemia or has BMI >= 30 kg/m2.
* Dyslipidemia was defined as having at least one of the following three conditions:

  * Low-density lipoprotein (LDL)-cholesterol level of > 3.4 mmol/L (> 130 mg/dL)
  * total cholesterol level of > 5.2 mmol/L (> 200 mg/dL)
  * triglyceride level of > 1.7 mmol/L (> 150 mg/dL). 254
* If the subject was female

  * she must either not of childbearing potential: defined as postmenopausal for at least 2 years or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy),
  * or was of childbearing potential and practicing one of the following methods of birth control: condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD)on contraceptives (oral or parenteral) for the 3-month period prior to Week 0, a vasectomized partner, total abstinence from sexual intercourse
* If the subject was female, the results of a urine pregnancy test performed at Screening and Week 0 were negative.
* If the subject was female, the subject was not breast-feeding.
* The subject was judged to be in general good health based upon the results of medical history, complete physical examination and clinical laboratory tests.
* The subject was not taking any over-the-counter or prescription drugs, or herbal products for weight loss during the 4 week period prior to Screening.
* The subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), prior to undertaking any study-specific procedures

Exclusion Criteria:

* History or evidence according to the 1997 American Diabetic Association (ADA)26criteria of type 1 or type 2 diabetes mellitus, i.e., fasting plasma glucose level >= 7.0 mmol/L.
* Inadequately controlled hypertension having systolic blood pressure >= 145 mmHg or diastolic blood pressure >= 90 mmHg (average of three measurements) or any hypertensive subjects taking > 3 medications to control blood pressure.
* History of Gilles de la Tourette's Syndrome.
* Use within 4 weeks prior to Week 0 of any of the following:

  * Monoamine oxidase inhibitors (MAOIs): used to treat depression and Parkinson's disease.
  * Medications that regulate the neurotransmitter serotonin in the brain (SSRIs): used to treat psychiatric disorders and to stop smoking.
  * Amino acids: used to treat sleep disorders.
  * Certain antimigraine drugs (such as sumatriptan, dihydroergotamine).
  * Opioids (such as pentazocine, pethidine, fentanyl, dextromethorphan).
* Organic causes of obesity (e.g., hypothyroidism).
* History of major eating disorders, such as anorexia nervosa or bulimia nervosa.
* History of benign prostatic hyperplasia with urinary retention.
* History of neurological disorders such as seizures.
* History of documented psychiatric illnesses such as anxiety, depression, bipolar disorder or schizophrenia or having psychotic symptoms.
* History or evidence of severe renal or hepatic impairments.
* History of narrow-angle glaucoma.
* History of coronary artery disease, congestive heart failure, peripheral arterial occlusive disease, arrhythmia or cerebrovascular disease (transient ischemic attacks or strokes).13. History or evidence of hyperthyroidism.
* Persistent tachycardia at rest, i.e., heart rate >100 bpm (average of 3 measurements).
* History of primary or secondary pulmonary hypertension.
* Underlying or suspected phaeochromocytoma.
* Known hypersensitivity to sibutramine hydrochloride monohydrate or any other component of the product.
* Known history of drug or alcohol abuse.
* Has previous history with the use of sibutramine.
* Any other medical illnesses judged by the investigator that may compromise the efficacy or safety of sibutramine.
* Unlikely to cooperate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2002-12; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Change in bodyweight from baseline to final evaluation | Wk 0, then, bi-weekly through duration of study

SECONDARY OUTCOMES:
The percentage of change in body weight from baseline to final evaluation. | Wk 0 and Wk 24
Total body fat mass, total body lean mass, percent of total body lean mass measurements (Bodystat® 1500) | Wks 0, 12 and 24
Total Abdominal Fat Mass, Total Abdominal Lean Mass, Percent of Total Abdominal Fat Mass and Percent of Total Abdominal Lean Mass (DEXA Scan) | Wk 0 and Wk 24
metabolic measurements (Cholesterol, Triglycerides & Insulin resistance) and SF 36 Quality of life measurement | Wk 0, 12 and Wk 24. In addition to the stated time frames, a Quality of life survey was conducted 30 days post study.